CLINICAL TRIAL: NCT05590728
Title: A Phase I, Open-label Study to Assess Lung Pharmacokinetics and Safety of a Single Dose of Apramycin Administered Intravenously in Healthy Adult Subjects
Brief Title: Safety of Intravenous Apramycin in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0012
Record Dates: First submitted 2022-07-21; First posted 2022-10-21 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2022-10-17

CONDITIONS: Bacterial Infection
Keywords: Apramycin; Lung Pharmacokinetics; Open-label; Phase I; Respiratory
MeSH Terms: conditions — Bacterial Infections | interventions — apramycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- T1 (Experimental): Subjects 18 to 45 years of age to receive 30 mg/kg apramycin dose administered intravenously (IV) in a forearm vein over 30 min (+/- 5 min) using a syringe or infusion pump. 0.5 h (+/- 5 min) after dosing a single bronchoscopy with bronchoalveolar lavage (BAL) will be performed to analyze concentration of apramycin in BAL. N=4
  Interventions: Drug: Apramycin (EBL-1003)
- T2 (Experimental): Subjects 18 to 45 years of age to receive single 30 mg/kg apramycin dose administered intravenously (IV) in a forearm vein over 30 min (+/- 5 min) using a syringe or infusion pump. 2 h (+/- 5 min) after dosing a single bronchoscopy with bronchoalveolar lavage (BAL) will be performed to analyze concentration of apramycin in BAL. N=4
  Interventions: Drug: Apramycin (EBL-1003)
- T3 (Experimental): Subjects 18 to 45 years of age to receive single 30 mg/kg apramycin dose administered intravenously (IV) in a forearm vein over 30 min (+/- 5 min) using a syringe or infusion pump. 4 h (+/-10 min) after dosing a single bronchoscopy with bronchoalveolar lavage (BAL) will be performed to analyze concentration of apramycin in BAL. N=4
  Interventions: Drug: Apramycin (EBL-1003)
- T4 (Experimental): Subjects 18 to 45 years of age to receive single 30 mg/kg apramycin dose administered intravenously (IV) in a forearm vein over 30 min (+/- 5 min) using a syringe or infusion pump. 8 h (+/- 15 min) after dosing a single bronchoscopy with bronchoalveolar lavage (BAL) will be performed to analyze concentration of apramycin in BAL. N=4
  Interventions: Drug: Apramycin (EBL-1003)
- T5 (Experimental): Subjects 18 to 45 years of age to receive single 30 mg/kg apramycin dose administered intravenously (IV) in a forearm vein over 30 min (+/- 5 min) using a syringe or infusion pump. Cohort T5 will be enrolled after plasma and lung apramycin concentrations and preliminary PK data analysis are completed in cohorts T1-T4 24 h (+/- 1 h) after dosing a single bronchoscopy with bronchoalveolar lavage (BAL) will be performed to analyze concentration of apramycin in BAL. N=4
  Interventions: Drug: Apramycin (EBL-1003)

INTERVENTIONS:
Drug: Apramycin (EBL-1003) — A mono-substituted 2-deoxystreptamine comprising a unique bicyclic octadiose moiety. It is a crystalline free base of the amoniglycoside apramycin.

SUMMARY:
A Phase I, open label study of a single dose of 30 mg/kg of apramycin administered intravenously (IV) over 30 (+/- 5) minutes. Twenty subjects will be enrolled in the study to one of 5 cohorts, T1-T5, each corresponding to a timepoint after initiation of infusion at which a single fiberoptic bronchoscopy with bronchoalveolar lavage (BAL) is performed. There will be 4 subjects per cohort. Cohort T5 will be enrolled after plasma and lung apramycin concentrations and preliminary PK data analysis are completed in cohorts T1-T4. Enrollment and dosing will be determined by bronchoscopy schedule. For each cohort, if 2 subjects are scheduled to receive study drug on the same day, the dose will be administered sequentially at least 2 hours apart. The primary objective is to assess plasma pharmacokinetic (PK) profile of apramycin and lung penetration of apramycin in epithelial lining fluid (ELF) and alveolar macrophages (AM) after single intravenous (IV) apramycin dose of 30 mg/kg in healthy subjects.

DETAILED DESCRIPTION:
A Phase I, open label study of a single dose of 30 mg/kg of apramycin administered intravenously (IV) over 30 (+/- 5) minutes. Twenty subjects will be enrolled in the study to one of 5 cohorts, T1-T5, each corresponding to a timepoint after initiation of infusion at which a single fiberoptic bronchoscopy with bronchoalveolar lavage (BAL) is performed. There will be 4 subjects per cohort. Cohort T5 will be enrolled after plasma and lung apramycin concentrations and preliminary PK data analysis are completed in cohorts T1-T4. Enrollment and dosing will be determined by bronchoscopy schedule. For each cohort, if 2 subjects are scheduled to receive study drug on the same day, the dose will be administered sequentially at least 2 hours apart. The primary objective is to assess plasma pharmacokinetic (PK) profile of apramycin and lung penetration of apramycin in epithelial lining fluid (ELF) and alveolar macrophages (AM) after single intravenous (IV) apramycin dose of 30 mg/kg in healthy subjects. The secondary objectives are to 1) assess the safety of single IV administration of 30 mg/kg apramycin in healthy subject and 2) to assess changes in otoacoustic testing.

ELIGIBILITY:
Inclusion Criteria:

1. Subject reads and signs the Informed Consent Form (ICF) and agree to have bronchoscopy with bronchoalveolar lavage under sedation or light anesthesia and comply with study procedures.
2. Healthy male or non-pregnant, non-lactating female subjects 18 to 45 years of age (both inclusive) at the time of dosing.

   *Note 1: Determined by medical history (MH), medication use, physical examination (PE), and vital signs, clinical laboratory tests and 12-lead ECG within reference ranges at Screening and Day-2. (See Sections 8.1 and 8.2; and Appendix B, Table 2, Table 3 and Table 4 and the study-specific MOP.)

   Exceptions to BP, HR and laboratory test values being with normal ranges are:
   * Abnormal HR and BP on first measurement may be repeated twice more with the subject resting between measurements for at least 5 min according to Section 8.1.6.
   * Subjects with baseline HR >/= 45 to 50 bpm may be accepted if otherwise healthy adults with known history of asymptomatic bradycardia.
   * Subjects with baseline SBP up to 140 mmHg and DBP up to 90 mmHg may be accepted if otherwise healthy.
   * A laboratory value that is Grade 1 will be allowed if not considered to be clinically significant by the investigator, with the exception of ALT, AST, AP, BUN, urine protein, serum creatinine or estimated glomerular filtration rate (eGFR) <70 mL/min /1.73 m^2 by the Chronic Kidney Disease Epidemiology collaboration (CKD-EPI) equation.
3. Female subjects of childbearing potential should use highly effective methods of contraception from the time of screening to 30 days after dosing.

   * Note 1: A female is considered of childbearing potential unless post-menopausal (defined as history of >/=1 year of spontaneous amenorrhea and a FSH level >40 IU/L), or permanently surgically sterilized.
   * Note 2: Highly effective contraceptive methods include: (a) surgical sterilization methods, such as tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful tubal obliteration (e.g., Essure(R)) with documented radiological confirmation test at least 90 days after the procedure, or (b) long-acting reversible contraception, such as progestin-releasing subdermal implants, copper intrauterine devices (IUDs), levonorgestrel-releasing IUDs.
   * Note 3: A subject who is not sexually active and abstains from sexual intercourse can be enrolled and abstinence documented.
4. Males, including vasectomized men, having sexual intercourse with women of childbearing potential must agree to consistent use of condoms from IMP administration through at least 30 days after dosing, and must also agree to not donate sperm during this same time period.

   *Note: A subject who is not sexually active and abstains from sexual intercourse can be enrolled and abstinence documented.
5. BMI 18.0 to 32.0 kg/m^2 (inclusive) and body weight not less than 50 kg.
6. Subjects with normal hearing, i.e., symmetric hearing with air conduction thresholds no worse than 20 dB hearing loss for the frequencies 0.5-1-2-4-6-8 kHz bilaterally.
7. Normal (reproducibility 70% or better) of distortion product otoacoustic emissions (DPOAEs).

   *Note: Absence of DPOAEs at no more than two consecutive or non-consecutive DPOAEs in each ear is acceptable.
8. Normal otoscopic findings in the ears, normal tympanic membrane mobility and stapedial reflex present.
9. From the signing of the informed consent until the last follow-up visit, subjects must be willing to avoid exposure to loud music or noise.

   *Note: Noise avoidance to include continuous usage of earpieces at high volume, attending loud concerts or dance events, or using firearms or attending fireworks.
10. Normal lung function with Forced Expiratory Volume in the first second (FEV1) predicted >/= 80% and FEV1/Forced Vital Capacity (FVC) > 70%.
11. Subjects must be willing to avoid excessive physical exercise within 48 h prior to dosing until discharge from the CTU on Day 3, and 24 h before each follow-up visit (Day 14 +/- 3 days and Day 30 +/- 4 days).
12. No history of acute febrile or infectious illness for at least 7 days prior to the administration of the IMP.
13. No history of lower respiratory tract infection within 4 weeks prior to screening.
14. Have adequate venous access for infusion and blood draws.

Exclusion Criteria:

All must be answered NO for the subject to be eligible for study participation:

1. Lactating females.

   Medical and surgical history:
2. Any history of hypersensitivity to aminoglycosides.
3. Any history of drug hypersensitivity, asthma, urticaria or other severe allergic diathesis.
4. Any history of seasonal allergies with ongoing symptoms for more than a week prior to dosing requiring glucocorticoids and/or frequent use of antihistamines for treatment.
5. Any history of a chronic condition that may increase risk to subject or interfere with endpoint assessment, or any unstable chronic disease.

   * Note 1: Unstable chronic disease is defined by need for frequent medical interventions that lead to a change in medications and/or required hospitalization, surgery or an invasive procedure or emergency department/urgent care visit.
   * Note 2: Any chronic disease, that has been diagnosed within 90 days of screening is excluded.
6. History of any psychiatric medical condition that has required hospitalization in the last 5 years or subject is considered psychologically unstable by the investigator.
7. History of acute or chronic problems with hearing and/or balance in the last 24 months.

   -Note: These include but not limited to use of hearing aid, head injury leading to otologic damage, tumor of the head or neck, autoimmune disease of the inner ear, tinnitus, vestibular disease, auditory neurinoma, endolymphatic hydrops and/or Meniere's disease, perilymphatic fistula, otitis media, labyrinthitis, sudden hearing loss, known retrocochlear hearing impairment, conductive hearing loss exceeding 10 dB at any frequency, ear canal and/or middle ear disease including inflammation or effusion, pathological tympanometry.
8. Past injury or surgery to the middle or inner ears.

   -Note: Myringotomy or tympanic tube insertion in childhood with complete healing and normal hearing test are excluded.
9. Family history of hearing loss before the age of 60.
10. Subjects who have had previous intolerance or contraindications to medications applied for sedation or anesthesia during bronchoscopy.

    -Note: These include benzodiazepines or topical anesthetic agents (lidocaine or xylocaine) including reversal agents such as flumazenil.

    Laboratory examinations:
11. Positive serum pregnancy test for women at screening or urine pregnancy test at check-in.
12. Positive test for HIV antibodies, hepatitis B-virus surface antigen (HBsAg), or anti-hepatitis C-virus antibodies (anti-HCV).

    Prior medication:
13. Use of any prescription or non-prescription medication prior to the dose of IMP

    -Note: Exceptions are hormonal contraceptives, which are permitted throughout the study, and solitary doses of up to 1,000 mg paracetamol.
14. Use of any investigational drug product within 30 days or 5 half-lives (whichever is longer) before dosing.
15. Planned participation in a clinical research study that requires treatment with a study drug or blood draws or other invasive assessments during the study period (screening until final visit).

    Lifestyle restrictions:
16. More than low-risk alcohol consumption (men: >/= 24 g of pure alcohol regularly per day; women: >/=12g of pure alcohol regularly per day) for the previous 3 months.
17. Any history of alcohol or drug abuse or positive alcohol breathalyzer test.
18. Suspicion of illicit drug use / abuse or positive urine drug screen test.
19. History of >/=10 pack-years smoking, or history of any nicotine use in the 6 months before check-in (Day -2) or positive urine cotinine screen at check-in.

    * Note 1: Nicotine products include cigarettes, e-cigarettes, pipe, cigar, chewing tobacco, nicotine patch.
    * Note 2: A positive urine cotinine at screening is allowed if negative at check-in (Day -2).
20. Caffeinated beverages/foods are prohibited within 48 hours before dosing to Day 3 of the trial. During the follow up period, consumption is restricted to not more than 3 cups or equivalent per day.
21. Judged by the investigator to have occupational noise exposure of high risk during the trial (e.g., construction site workers, military workers, etc.).
22. Blood or plasma donation of 500 mL within 3 months or more than 100 mL within 30 days before signing informed consent or planned donation prior to completion of this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alliance for Multispecialty Research, LLC - Knoxville, Knoxville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included healthy male and female adults, ages 18-45 years, inclusive, who met all eligibility criteria. Participants were enrolled between May 15, 2023 and October 16, 2023 and were recruited from the community at large.
Pre-assignment Details: Participants who signed the Informed Consent Form underwent screening procedures that included medical history, physical exam, clinical laboratory testing (hematology, chemistry, coagulation, urinalysis, viral serology (for HIV, HCV and HBV), and pregnancy testing. Participants who met all the inclusion criteria and none of the exclusion criteria were admitted into the clinical trial unit to confirm eligibility on Day -1 and assigned to one of the study cohorts before dosing on Day 1.
Groups:
- 30 Minute BAL: A single 30 mg/kg apramycin dose was administered intravenously (IV) in a total volume of 30 mL over 30 minutes (+/- 5 minutes) to each participant. Bronchoscopy with bronchoalveolar lavage (BAL) performed 30 minutes (+/- 5 minutes) after infusion start.
  Apramycin (EBL-1003): A mono-substituted 2- deoxystreptamine comprising a unique bicyclic octadiose moiety. It is a crystalline free base of the aminoglycoside apramycin. Apramycin for infusion is formulated as 150 mg free base /mL in sterile aqueous solution, pH 5.5 to 6.0 adjusted with sulfuric acid. The study product is supplied in 20 mL glass vials. Based on the participant's weight, the appropriate weight-based apramycin for infusion dose was calculated and the appropriate number of vials were removed from storage to prepare the infusion. Sterile normal saline was used to adjust the infusion volume.
- 2 Hour BAL: A single 30 mg/kg apramycin dose was administered intravenously (IV) in a total volume of 30 mL over 30 minutes (+/- 5 minutes) to each participant. Bronchoscopy with bronchoalveolar lavage (BAL) performed 2 hours (+/- 5 minutes) after infusion start.
  Apramycin (EBL-1003): A mono-substituted 2- deoxystreptamine comprising a unique bicyclic octadiose moiety. It is a crystalline free base of the aminoglycoside apramycin. Apramycin for infusion is formulated as 150 mg free base /mL in sterile aqueous solution, pH 5.5 to 6.0 adjusted with sulfuric acid. The study product is supplied in 20 mL glass vials. Based on the participant's weight, the appropriate weight-based apramycin for infusion dose was calculated and the appropriate number of vials were removed from storage to prepare the infusion. Sterile normal saline was used to adjust the infusion volume.
- 4 Hour BAL: A single 30 mg/kg apramycin dose was administered intravenously (IV) in a total volume of 30 mL over 30 minutes (+/- 5 minutes) to each participant. Bronchoscopy with bronchoalveolar lavage (BAL) performed 4 hours (+/- 10 minutes) after infusion start.
  Apramycin (EBL-1003): A mono-substituted 2- deoxystreptamine comprising a unique bicyclic octadiose moiety. It is a crystalline free base of the aminoglycoside apramycin. Apramycin for infusion is formulated as 150 mg free base /mL in sterile aqueous solution, pH 5.5 to 6.0 adjusted with sulfuric acid. The study product is supplied in 20 mL glass vials. Based on the participant's weight, the appropriate weight-based apramycin for infusion dose was calculated and the appropriate number of vials were removed from storage to prepare the infusion. Sterile normal saline was used to adjust the infusion volume.
- 8 Hour BAL: A single 30 mg/kg apramycin dose was administered intravenously (IV) in a total volume of 30 mL over 30 minutes (+/- 5 minutes) to each participant. Bronchoscopy with bronchoalveolar lavage (BAL) performed 8 hours (+/- 15 minutes) after infusion start.
  Apramycin (EBL-1003): A mono-substituted 2- deoxystreptamine comprising a unique bicyclic octadiose moiety. It is a crystalline free base of the aminoglycoside apramycin. Apramycin for infusion is formulated as 150 mg free base /mL in sterile aqueous solution, pH 5.5 to 6.0 adjusted with sulfuric acid. The study product is supplied in 20 mL glass vials. Based on the participant's weight, the appropriate weight-based apramycin for infusion dose was calculated and the appropriate number of vials were removed from storage to prepare the infusion. Sterile normal saline was used to adjust the infusion volume.
- 24 Hour BAL: A single 30 mg/kg apramycin dose was administered intravenously (IV) in a total volume of 30 mL over 30 minutes (+/- 5 minutes) to each participant. Bronchoscopy with bronchoalveolar lavage (BAL) performed 24 hours (+/- 1 hours) after infusion start. This cohort was not enrolled due to hearing impairment adverse events (AEs) experienced by participants in the first 4 cohorts.
  Apramycin (EBL-1003): A mono-substituted 2- deoxystreptamine comprising a unique bicyclic octadiose moiety. It is a crystalline free base of the aminoglycoside apramycin. Apramycin for infusion is formulated as 150 mg free base /mL in sterile aqueous solution, pH 5.5 to 6.0 adjusted with sulfuric acid. The study product is supplied in 20 mL glass vials. Based on the participant's weight, the appropriate weight-based apramycin for infusion dose was calculated and the appropriate number of vials were removed from storage to prepare the infusion. Sterile normal saline was used to adjust the infusion volume.
Period: Overall Study
Arm/Group | 30 Minute BAL | 2 Hour BAL | 4 Hour BAL | 8 Hour BAL | 24 Hour BAL
Started | 4 | 4 | 4 | 4 | 0
Started Infusion | 4 | 4 | 4 | 4 | 0
Completed Infusion | 4 | 4 | 4 | 4 | 0
Completed Bronchoscopy With BAL | 4 | 4 | 4 | 4 | 0
Completed All PK Blood Draws | 3 | 4 | 4 | 4 | 0
Completed All Plasma Urea Blood Draws | 3 | 4 | 4 | 4 | 0
Completed | 4 | 4 | 4 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population includes all participants who received any amount of apramycin.
Groups:
- Total: Total of all reporting groups
Arm/Group | 30 Minute BAL | 2 Hour BAL | 4 Hour BAL | 8 Hour BAL | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (10.0) | 34.0 (3.5) | 27.0 (6.2) | 30.5 (8.8) | 30.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4 | 8
  Male | 2 | 3 | 3 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 4 | 4 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 2 | 0 | 4
  White | 3 | 2 | 2 | 3 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.13 (2.70) | 27.08 (2.84) | 24.50 (3.28) | 26.78 (3.10) | 26.62 (3.00)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to 8 h (AUC 0-8) of Total Apramycin in Epithelial Lining Fluid (ELF) and Alveolar Macrophage (AM)
Description: AUC 0-8 (ug*h/mL) was estimated using Phoenix WinNonlin Non-compartmental analysis. Each participant only contributed one ELF and AM concentration at one time point, so the PK parameters for ELF and AM were calculated using the geometric mean (GM) concentration at each BAL sampling time point, resulting in a single parameter estimate of ELF and AM across all participants.
Time Frame: 0 h through 8 h post dose
Population: The PK Analysis Subset population includes all participants who completed the lung and plasma PK parts of the trial without any protocol deviations that would likely affect the PK results and who have evaluable plasma PK and BAL PK concentration data for apramycin. All cohorts are reported jointly as all received the same dose, following the same dosing schedule.
Measure: Number; unit: ug*h/mL
Groups:
- Apramycin All Participants: A single 30 mg/kg apramycin dose administered intravenously (IV) over 30 minutes (+/- 5 minutes).
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 11
ug*h/mL
  ELF | 142.8
  AM | 131.7

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC 0-inf) of Total Apramycin in ELF and AM
Description: AUC 0-inf (ug*h/mL) was estimated using Phoenix WinNonlin Non-compartmental analysis. Each participant only contributed one ELF and AM concentration at one time point, so the PK parameters for ELF and AM were calculated using the geometric mean (GM) concentration at each BAL sampling time point, resulting in a single parameter estimate of ELF and AM across all participants.
Time Frame: 0 h through 8 h post dose
Population: as for outcome 1
Measure: Number; unit: ug*h/mL
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 11
ug*h/mL
  ELF | 197.3
  AM | NA — Phoenix WinNonlin could not calculate an estimate for this PK parameter.

3. Primary Outcome: Maximum Concentration (Cmax) of Total Apramycin in ELF and AM
Description: Cmax (ug/mL) was estimated using Phoenix WinNonlin Non-compartmental analysis. Each participant only contributed one ELF and AM concentration at one time point, so the PK parameters for ELF and AM were calculated using the geometric mean (GM) concentration at each BAL sampling time point, resulting in a single parameter estimate of ELF and AM across all participants.
Time Frame: 0 h though 8 h post dose
Population: as for outcome 1
Measure: Number; unit: ug/mL
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 11
ug/mL
  ELF | 27.47
  AM | 42.37

4. Primary Outcome: Time of Maximum Concentration (Tmax) of Total Apramycin in ELF and AM
Description: Tmax (h) was estimated using Phoenix WinNonlin Non-compartmental analysis. Each participant only contributed one ELF and AM concentration at one time point, so the PK parameters for ELF and AM were calculated using the geometric mean (GM) concentration at each BAL sampling time point, resulting in a single parameter estimate of ELF and AM across all participants.
Time Frame: 0 h through 8 h post dose
Population: as for outcome 1
Measure: Number; unit: h
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 11
h
  ELF | 0.5
  AM | 8

5. Primary Outcome: Terminal Elimination Half-Life (t1/2) of Total Apramycin in ELF and AM
Description: t1/2 (h) was estimated using Phoenix WinNonlin Non-compartmental analysis. Each participant only contributed one ELF and AM concentration at one time point, so the PK parameters for ELF and AM were calculated using the geometric mean (GM) concentration at each BAL sampling time point, resulting in a single parameter estimate of ELF and AM across all participants.
Time Frame: 0 h through 8 h post dose
Population: as for outcome 1
Measure: Number; unit: h
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 11
h
  ELF | 4.05
  AM | NA — Phoenix WinNonlin could not calculate an estimate for this PK parameter.

6. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to 8 h (AUC 0-8) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of AUC 0-8 (h*ug/mL). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study.
Time Frame: 0 h through 8 h post dose
Population: The Plasma PK population consists of all participants who received a complete dose of apramycin and have at least one quantifiable post-dose plasma drug concentration measured. All cohorts are reported jointly as all received the same dose, following the same dosing schedule.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
ug*h/mL | 443.9 (11)

7. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 h (AUC 0-24) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of AUC 0-24 (h*ug/mL). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study.
Time Frame: 0 h through 24 h post dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
ug*h/mL | 486.7 (13)

8. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Measurable Concentration Above the Lower Limit of Quantitation (AUC 0-last) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of AUC (0-last) (h*µg/mL). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study.
Time Frame: 0 h through 60 h post dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
ug*h/mL | 490.3 (13)

9. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC 0-inf) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of AUC (0-Inf) (h*µg/mL). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study. AUC 0-Inf was estimated for plasma concentration data with the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) = 0.90 and includes at least 3 timepoints after time to maximum concentration (Tmax).
Time Frame: 0 h through 60 h post dose
Population: The Plasma PK population consists of all participants who received a complete dose of apramycin and have at least one quantifiable post-dose plasma drug concentration measured. All cohorts are reported jointly as all received the same dose, following the same dosing schedule. Four participants' concentration data did not meet the lambda-z acceptance criteria and are not included in the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/mL
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 12
ug*h/mL | 500.3 (14)

10. Primary Outcome: Maximum Concentration (Cmax) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of Cmax (ug/mL). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study.
Time Frame: 0 h though 60 h post dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
ug/mL | 172.1 (10)

11. Primary Outcome: Time of Maximum Concentration (Tmax) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of Tmax (h). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study.
Time Frame: 0 h through 60 h post dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
h | 0.595 (32)

12. Primary Outcome: Terminal Elimination Half-Life (t1/2) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of t1/2 (h). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study. t1/2 was estimated for plasma concentration data with the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) = 0.90 and includes at least 3 timepoints after time to maximum concentration (Tmax).
Time Frame: 0 h through 60 h post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 12
h | 19.1 (19)

13. Primary Outcome: Central Volume of Distribution (Vd) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of Vd (L/kg). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study. Vd was estimated for plasma concentration data with the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) = 0.90 and includes at least 3 timepoints after time to maximum concentration (Tmax).
Time Frame: 0 h to 60 h post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 12
L/kg | 1.64 (22)

14. Primary Outcome: Total Clearance (CLT) of Total Apramycin in Plasma
Description: Geometric mean (GM) and coefficient of variation as a percent (CV%) of CLT (L/h/kg). PK parameters were estimated from the total apramycin plasma concentration-time data after a complete dose using Phoenix WinNonlin Non-compartmental analysis. Plasma concentrations were measured by a validated LC-MC/MS bioanalytical assay for plasma samples collected during the study. CLT was estimated for plasma concentration data with the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) = 0.90 and includes at least 3 timepoints after time to maximum concentration (Tmax).
Time Frame: 0 h through 60 h post dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/kg
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 12
L/h/kg | 0.0600 (14)

15. Primary Outcome: Ratio of ELF to Plasma and AM to Plasma Apramycin Exposure Parameters
Description: The ratios for Cmax (ug/mL), AUC 0-8 (ug*h/mL), and AUC 0-inf (ug*h/mL) of ELF to plasma and AM to plasma were calculated by dividing the Cmax (ug/mL), AUC 0-8 (ug*h/mL), and AUC 0-inf (ug*h/mL) of ELF and AM by the Cmax (ug/mL), AUC 0-8 (ug*h/mL), and AUC 0-inf (ug*h/mL) of total apramycin in plasma, respectively. All PK parameters were estimated using Phoenix WinNonlin Non-compartmental analysis. Each participant only contributed one ELF and AM concentration at one time point, so the PK parameters for ELF and AM were calculated using the GM concentration at each BAL sampling time point, resulting in a single parameter estimate of ELF and AM across all participants. The PK parameters for total apramycin in plasma were calculated using the GM result of the total apramycin in plasma concentrations at the corresponding BAL time point.
Time Frame: 0 h through 8 h post dose
Population: as for outcome 1
Measure: Number; unit: ratio of lung PK to plasma PK
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 11
ratio of lung PK to plasma PK
  Cmax, ELF to Plasma | 0.144
  Cmax, AM to Plasma | 0.222
  AUC 0-8, ELF to Plasma | 0.324
  AUC 0-8, AM to Plasma | 0.299
  AUC 0-inf, ELF to Plasma | 0.404
  AUC 0-inf, AM to Plasma | NA — Phoenix WinNonlin could not calculate an estimate of AUC 0-inf for AM, so a ratio could not be calculated.

16. Secondary Outcome: Frequency of Serious Adverse Events (SAEs)
Description: Number of participants that experience any SAEs from Day 1 to Day 30. An AE is considered serious if, in the view of either the site principal investigator or sponsor, it results in: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 30
Population: The safety population includes all participants who received any amount of apramycin. All participants received the same dose of study product and are therefore reported jointly for safety outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants | 0

17. Secondary Outcome: Frequency of Treatment-emergent Adverse Events (TEAEs)
Description: The number of participants who experienced at least one unsolicited TEAE of any severity and relatedness. Any medical condition that was present at screening was considered a baseline finding and not reported as an AE. However, if the grade increased at any time during the trial such that it met the AE definition, it was recorded as an AE.
Time Frame: Day 1 through Day 30
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants
  Ear and labyrinth disorders | 4
  Eye disorders | 1
  General disorders and administration site conditions | 1
  Infections and infestations | 1
  Injury, poisoning and procedural complications | 1
  Investigations | 5
  Nervous system disorders | 1
  Respiratory, thoracic and mediastinal disorders | 2

18. Secondary Outcome: Frequency of Abnormal Physical Exam Findings
Description: Abnormal physical exam findings through Day 14. Physical exams included assessment of head, eyes, ears, nose, and throat; heart, lungs, abdomen, skin, musculoskeletal system, and lymph nodes.
Time Frame: Day 1 through Day 14
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants
  Head, Eyes, Ears, Nose, Throat (HEENT) | 2
  Musculoskeletal | 1

19. Secondary Outcome: Frequency of Abnormal Vital Sign Findings
Description: Abnormal vital sign findings through Day 14. Vital sign measurements include systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, and oral temperature. If a vital sign finding met the threshold for an AE at baseline, subsequent vital sign results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 14
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants
  Systolic blood pressure - decrease | 1
  Systolic blood pressure - increase | 0
  Diastolic blood pressure - decrease | 0
  Diastolic blood pressure - increase | 0
  Pulse - decrease | 2
  Pulse - increase | 0
  Respiratory rate - decrease | 0
  Respiratory rate - increase | 0
  Oral temperature - decrease | 0
  Oral temperature - increase | 5

20. Secondary Outcome: Frequency of Abnormal Chemistry Lab Measurements
Description: Abnormal chemistry laboratory findings through Day 14. Graded chemistry laboratory measurements include sodium, potassium, glucose (fasting), blood urea nitrogen, creatinine, calcium, magnesium, carbon dioxide, albumin, total protein, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, total bilirubin, and direct bilirubin. If a clinical chemistry laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 14
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants
  Sodium - decrease | 0
  Sodium - increase | 0
  Potassium - decrease | 0
  Potassium - increase | 0
  Glucose - decrease | 0
  Glucose - increase | 2
  Blood urea nitrogen - increase | 0
  Creatinine - increase | 0
  Calcium - decrease | 0
  Calcium - increase | 1
  Magnesium - decrease | 0
  Carbon dioxide - decrease | 0
  Carbon dioxide - increase | 3
  Albumin - decrease | 1
  Total protein - decrease | 0
  Alkaline phosphatase - increase | 0
  Alanine aminotransferase - increase | 0
  Aspartate aminotransferase - increase | 0
  Total bilirubin - increase | 1
  Direct bilirubin - increase | 0

21. Secondary Outcome: Frequency of Abnormal Hematology Lab Measurements
Description: Abnormal hematology laboratory findings through Day 14. Graded hematology laboratory measurements include hemoglobin, platelet count, white blood cells, neutrophils, lymphocytes, eosinophils, basophils, and monocytes. If a clinical hematology laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 14
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants
  Hemoglobin - decrease | 0
  Platelets - decrease | 0
  White blood cells - decrease | 2
  White blood cells - increase | 2
  Neutrophils - decrease | 0
  Lymphocytes - decrease | 0
  Eosinophils - increase | 1
  Basophils - increase | 0
  Monocytes - increase | 1

22. Secondary Outcome: Frequency of Abnormal Coagulation Lab Measurements
Description: Abnormal coagulation laboratory findings through Day 14. Graded coagulation laboratory measurements include activated partial thromboplastin time, prothrombin time, and prothrombin international normalized ratio. If a clinical coagulation laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 14
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants
  Activated partial thromboplastin time - increase | 3
  Prothrombin time - increase | 2
  Prothrombin international normalized ratio - increase | 2

23. Secondary Outcome: Frequency of Abnormal Urinalysis Lab Measurements
Description: Abnormal urinalysis laboratory findings through Day 14. Urinalysis laboratory measurements include routine dipstick testing of clean-catch urine for blood, protein, and glucose. If urine dipstick was abnormal, urine microscopy was performed. If a clinical urinalysis laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 14
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants
  Protein by dipstick - increase | 2
  Glucose by dipstick - increase | 0
  Blood by dipstick - increase | 4
  White blood cells by microscopy - increase: number analyzed (Participants) | 11
  White blood cells by microscopy - increase | 0
  Red blood cells by microscopy - increase: number analyzed (Participants) | 11
  Red blood cells by microscopy - increase | 1
  Bacteria by microscopy - increase: number analyzed (Participants) | 11
  Bacteria by microscopy - increase | 1

24. Secondary Outcome: Frequency of Abnormal Changes in Electrocardiographic (ECG) Results
Description: Changes in ECG intervals and morphological changes from baseline up to 24 hours after dosing. The graded ECG measurements include PR interval and QTcF interval.
Time Frame: 0 h through 24 h post dose
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants
  PR interval | 0
  QTcF interval | 0

25. Secondary Outcome: Frequency of Audiology TEAEs
Description: TEAEs related to auditory (cochlear) function tests (pure-tone audiometry and distortion product otoacoustic emissions [DPOAEs]) through Day 30.
Time Frame: Day 1 through Day 30
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Apramycin All Participants
Number analyzed (Participants) | 16
Participants | 4

ADVERSE EVENTS:
Time Frame: All treatment emergent adverse events (TEAEs) were documented from time of study drug dosing through the time of last assessment (e.g., Day 14 +/- 3 days of clinical safety labs and ECGs) or Final Visit (Day 30 +/- 4 days).
Description: Any systemic medical condition, vital sign and ECG measurement, and clinical safety lab test value that was present on Day 1 prior to dosing was considered a baseline finding. For ear and otoacoustic testing, baseline comprises of assessment performed on Day -2. If the condition increases in severity or frequency after study product administration, it was reported as a TEAE. All participants received the same dose of study product and are therefore jointly reported for adverse events.
Arm/Group | Apramycin All Participants
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apramycin All Participants (N=16)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 4 (5)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure systolic decreased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 3 (4)
Heart rate decreased (Investigations) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3)
Bacterial test positive (Investigations) | 1 (1)
Bilirubin conjugated increased (Investigations) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1)
Blood calcium increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 2 (2)
Blood urine present (Investigations) | 4 (4)
Carbon dioxide increased (Investigations) | 3 (3)
Eosinophil count increased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 2 (2)
Monocyte count increased (Investigations) | 1 (1)
Protein urine present (Investigations) | 2 (2)
Prothrombin time prolonged (Investigations) | 2 (2)
Red blood cells urine positive (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2)
White blood cell count increased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT05590728/Prot_001.pdf
  • Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT05590728/SAP_002.pdf
  • Informed Consent Form (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT05590728/ICF_000.pdf